CLINICAL TRIAL: NCT05358093
Title: Retrospective Study of Cardiac Toxicity of Hypo Fractionated Radiotherapy in Left Breast Cancer
Brief Title: Cardiac Toxicity of Hypo Fractionated Radiotherapy in Left Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Hussien Ahmed Hussien, principle investigator, Assiut University
Other Study IDs: left breast cancer
Record Dates: First submitted 2022-03-30; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 45

SUMMARY:
Worldwide, Breast cancer is the most common cancer in women,where 1.7 million new cases diagnosed in 2012 . In 2020 number doubled as 2.3 million women diagnosed with breast cancer. According to ACS 1 in 8 women in United states will develop breast cancer in her life .

Similarly again, In Egypt breast cancer is the most common malignancy in women about 22,700 new cases recorded in 2020. Accounting for 38.8% of cancers in this population and forecasted to be approximately 46,000 in 2050 .

Post-operative radiotherapy is fundamental part of treatment after either conservative surgery or mastectomy . Conventionally fractionated radiation therapy (CFRT) ,Delivering 45-50 GY in 1.8-2 GY daily fractions for 5 days per week over 5-7 weeks was the standard schedule to eradicate sub clinical disease ,sparing normal tissues .After the publication of long term results of randomized controlled trials (RCTs) comparing safety and effectiveness of hypo fractionated RT (HFRT)delivered in3 weeks ,vs. CFRT in node negative BC has been implemented . in 2008 numerous international guidelines recommended HFRT as the new standard being Cost effectiveness ,limited resources ,excessively long RT waiting lists ,Another important argument for HFRT utilization ,even assuming alpha/beta of 1.5GY ,is biologically milder or isoeffective for healthy tissues compered to CFRT .

Cardiac toxicity is potentially long or short term complication of various anticancer therapies systemic therapy as anthracyclines or biological agent implicated in causing irreversible cardiac dysfunction.

Radiotherapy also have cardio toxic effect through different mechanisms

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years old 2. histopathology diagnosed 3. Left sided breast cancer 4. Receiving 3D hypofractionated radiotherapy 5. Patients should be non metastatic 6. performance status 0-2

Exclusion Criteria:

* • Patient > 75 years old

  * Non histological diagnosed
  * Metastatic patient
  * Patient with cardiac or other co morbidity.
  * ECoG performance status >2
  * pregnant or lactating patients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female with left breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-04-27 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
retrospective study of cardiac toxicity in left breast cancer received hypofractionated radiotherapy | baseline
  detection of toxicity on cardiac ejection fraction in 45 patients received hypofractionated radiotherapy over left breast

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://seer.cancer.gov/csr/1975_2012/
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/12165639